CLINICAL TRIAL: NCT04864145
Title: Transcatheter Self-expandable Valve Implantation for the Treatment of Severe Native Aortic Regurgitation: a Prospective, Multicenter, Randomized Study
Brief Title: Transcatheter Self-expandable Valve Implantation for the Treatment of Severe Native Aortic Regurgitation
Acronym: SEASON-AR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Director of Cardiology and Cath Lab, Vice President of Nanjing First Hospital, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20210325
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement; Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical therapy (Active Comparator): Patients in medical therapy will receive conservative care, mainly including angiotensin-neprilysin inhibition (ARNI), diuretics, dihydropyridine calcium channel blocker, angiotensin-converting enzyme (ACE) inhibitors/angiotensin receptor blockers (ARBs) or beta blockers.
  Interventions: Drug: Medical therapy
- Transcatheter Aortic Valve Implantation (Experimental): Patients in TAVR group will receive transcatheter aortic valve replacement.
  Interventions: Device: Transcatheter Aortic Valve Implantation

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation — The VitaFlow™ system (MicroPort®, Shanghai, China) was a novel TAVR system, which incorporates high-radial force and a double layer polyethylene terephthalate (PET) skirt to optimize frame geometry and minimize the risks of paravalvular leak (PVL). The VitaFlow™ transcatheter aortic valve is made of a self-expanding nitinol frame and tri-leaflet bovine pericardial valve.
  Other Names: The VitaFlow™ system (MicroPort®, Shanghai, China)
  Arms: Transcatheter Aortic Valve Implantation
Drug: Medical therapy — Angiotensin-neprilysin inhibition (ARNI), diuretics, dihydropyridine calcium channel blocker, angiotensin-converting enzyme (ACE) inhibitors/angiotensin receptor blockers (ARBs) or beta blockers.
  Other Names: Optimal medical therapy
  Arms: Medical therapy

SUMMARY:
Prospective, multicenter, randomized trial.

DETAILED DESCRIPTION:
Patients with severe native aortic valve regurgitation (AR) who have symptoms, impaired LVEF (≤55%) or left ventricular enlargement have the indications for surgery. According to data from the Euro Heart Survey, only 21.8% with LVEF 30-50% and 2.7% with LVEF <30% were referred for surgical aortic valve replacement (SAVR) among patients with severe native aortic regurgitation. Advanced age and comorbidities were often considered as main reasons to refuse SAVR. The annual mortality of untreated patients with severe AR is 10-20%. Pure native AR is always an exclusion criterion in all randomized controlled trials on transcatheter aortic valve implantation (TAVR) because the specific anatomical features can preclude adequate valve implantation. Several small, retrospective studies showed that off-label use of TAVR appears to be a feasible treatment choice for AR patients at high risk for SAVR. The present study aims to investigate the use of TAVR in AR patients.

ELIGIBILITY:
Inclusion Criteria:

1. Procedural indications: symptomatic severe aortic regurgitation; no symptom plus left ventricular ejection fraction ≤ 55% or left ventricular end-diastolic dimension (LVEDD) > 65mm or left ventricular end-systolic dimension (LVESD) > 50mm;
2. Severe aortic valve regurgitation, and mean pressure gradient < 20mmHg; Annular perimeter ≤ 85 mm;
3. The ratio of the perimeter of the left ventricular outflow tract 4mm to the perimeter of the valve annulus is 0.95-1.05;
4. STS score ≥8 or moderate to severe frailty or refused surgical valve replacement or presence of any of the following factors judged to be difficult to perform the surgical valve replacement:

   1. Severe aorta calcification or active ascending aorta atherosclerotic plaque
   2. History of mediastinum radiotherapy
   3. Past mediastinitis
   4. Presence of unobstructed coronary bypass implants
   5. Previous more than two cardiothoracic surgeries
   6. Liver cirrhosis
   7. Other surgical risk factors

Exclusion Criteria:

1. Age < 60 years old;
2. Ascending aorta diameter >45mm;
3. Coronary multi-vessel disease (SYNTAX score >32);
4. Life expectancy <1 year;
5. Left ventricular ejection fraction <30%;
6. Acute myocardial infarction within 30 days;
7. Allergies or contraindications to related drugs (aspirin, clopidogrel, warfarin, or contrast agents);
8. Other situations judged by the researcher as unsuitable for participating in the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinical worsening | 12 months
  A composite of all cause death, disabling stroke, or heart failure rehospitalization

SECONDARY OUTCOMES:
Procedural complications | 12 months
  Any aortic dissection, annular rupture, coronary artery occlusion, vascular complications, permanent pacemaker implantation.
6-minute walk distance | 12 months
  This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes.
New York Heart Association (NYHA) functional class | 12 months
  Classification of function capacity of the NYHA.
Stroke | 12 months
  Stroke is defined as an acute episode of focal or global neurological dysfunction caused by the brain, spinal cord, or retinal vascular injury as a result of hemorrhage or infarction.
Mortality | 12 months
  All-cause, cardiovascular, and non-cardiovascular mortality
Bleeding Complications | 12 months
  The original VARC definitions with BARC classifications
Prothetic valve dysfunction | 12 months
  Any prothetic aortic valve stenosis, prothesis-patient mismatch, prosthetic aortic valve regurgitation
Rehospitalization | 12 months
  Requiring hospitalizations for valve-related symptoms or worsening congestive heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China